CLINICAL TRIAL: NCT06108661
Title: Effects of ELDOA and Slump Stretching on Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/21
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial which will consist of two groups. Once will receive conventional physical therapy and the second will receive conventional physical therapy and slump stretching. Both groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be a another person who will be unaware of the group the participant belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Treatment protocol given to both groups will be carried out for 3 sessions per week for 2 weeks.
  It will comprise of hot pack for 10 minutes in prone position. Stretching protocol for shortened muscles. Frequency would be: 3 times per week (alternatively) for 1st week and 2nd week.
  ELDOA. As per the tolerance of the patient. (Max hold time=60sec) For 2 weeks (alternatively).
  Interventions: Procedure: Conventional Physical Therapy; Procedure: ELDOA
- Group B (Active Comparator): Treatment protocol given to both groups will be carried out for 3 sessions per week for 2 weeks.
  It will comprise of hot pack for 10 minutes. Stretching protocol for shortened muscles. Frequency would be: 3 times per week (alternatively) for 1st week and 2nd week.
  Slump Stretching: Slump stretching will be performed with the patient in the long sitting position with the patient's feet against the wall to assure the ankle remained in 0 degree dorsiflexion. The therapist will apply over pressure to the cervical spine flexion to the point where the patient's symptoms will be reproduced. The position will be held for 30 s. A total of 5 repetitions will be completed
  Interventions: Procedure: Conventional Physical Therapy; Procedure: Slump Stretching

INTERVENTIONS:
Procedure: Conventional Physical Therapy — Moist heat therapy for 10 minutes for 3 times per week (alternatively) for 2 weeks.
  TENS was applied for 15 minutes, 3 times per week (alternatively) for 2 weeks. Stretching protocol for deep lumbar spinal muscles was employed. The frequency was 3 times per week (alternatively) for 2 weeks.
Procedure: Slump Stretching — Slump stretching will be performed with the patient in the long sitting position with the patient's feet against the wall to assure the ankle remained in 0 degree dorsiflexion. The therapist will apply over pressure to the cervical spine flexion to the point where the patient's symptoms will be reproduced. The position will be held for 30 s. A total of 5 repetitions will be completed.
  Arms: Group B
Procedure: ELDOA — ELDOA will be performed as per the tolerance of the patient (Max hold time=60sec) for 2 weeks (alternatively). For L4/L5 spinal segment patient sits on the floor, arms at the side legs relaxed.
  For L5/S1 segment the patient lies on his or her side with torso perpendicular to a wall with the sitz bone pressing into the wall. The patient swing the legs up so that he or she is lying on his or her back with the legs perpendicular up the wall and the sitz bone pressing into the wall. The arms are lying by the sides.
  Arms: Group A

SUMMARY:
The title of this study is Shirt term effects of ELDOA and slump steyching in mechanical low back pain. Previous studies have identified the effects of ELDOA and slump stretching on mechanical low back pain, but their short term effects have not been compared. This study will focus on the comparison of these techniques and their effectiveness in patients with mechanical low back pain. The purpose of this study is to compare the short term effects of ELDOA and slump stretching on spatiotemporal gait parameters, lumbar ROM and pain in patients with mechanical low back pain.

Spatiotemporal gait parameters will be measured by using formulas. Participants of interest would be approached and explained about the research. Informed written consent will be taken. Recruited participants will be allocated to either of the groups through a sealed opaque envelope method. ELODA and slump stretching will be given to groups A and B respectively, along with conventional physical therapy treatment. Inclinometer, NPRS and formulas for spatiotemporal gait parameters will be used as outcome measures.

DETAILED DESCRIPTION:
Low back pain is one of the most prevalent musculoskeletal conditions worldwide. Amongst the general population, more than 70% of the people experience low back pain at some time in their lifetime. The prevalence of low back pain was found to be 32%,52%,96%,72.8 %,72.9%, 56.6%,56.25%, 69 % in school teachers, bankers, dentists, nurses, clinical physical therapist, health science students, Salesmen and computer users respectively in Pakistan. Low back pain is pain or discomfort in the lumbosacral region from the lower costal margin to the inferior gluteal fold.

This randomized control trial will be conducted in MDL2 of Foundation University College of Physical Therapy using non-probability purposive sampling. Participants will be briefed regarding the study objectives, procedure, risks and benefits of treament, voluntary participation and right to withdraw. Written informed consent will be taken from all the participants before conducting the research. Details of exercise program will be explained to them. Diagnostic tests will be applied to confirm the Low back pain. Slump test will be used for this purpose. Then the selected participants will be randomized into 2 groups(experimental group and control group)via lottery method. Participants will complete Numeric Rating Pain Scale(NRPS) for pain. Lumbar ROM and spatiotemporal gait parameters will be noted. All of these measurements will be taken at baseline, after 1 week and then after 2 weeks of intervention.

The treatment protocol of both groups is as follows:

Group 1(Experimental group): Conservative management including hot pack, TENS and muscle stretching along with ELDOA (each position will be maintained as per the tolerance of the patient).

Group 2(Control group): Conservative management including hot pack, TENS and muscle stretching along with slump stretching (position will be maintained as per the tolerance of the patient).

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-45 years old
* Both males and females
* Patients with pain intensity of at least 5 on NPRS
* Positive slump test

Exclusion Criteria:

* Any congenital deformities
* Demonstrated neurological deficit
* Pregnant females
* History of spinal surgery
* Spondylolisthesis
* Severe lumbar spondylosis
* Spinal stenosis
* Disc herniation
* Serious spinal conditions like infection, tumors, osteoporosis, spinal fracture
* Limb length discrepancy
* Sacroiliac and hip disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-12-05 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Lumbar ROM | 2 weeks
  Inclinometer will be used to measure the lumbar ROM. One inclinometer is placed on T12 spinous process and the second inclinometer is placed on S1 spinous process of participant. The patient is asked to perform forward flexion, extension and lateral flexion, The range of motion is recorded by subtracting the value on lower inclinometer from upper inclinometer
Gait speed: | 2 weeks
  Gait speed = distance(m) x time(s)
Cycle time | 2 weeks
  Cycle time(s) = time(s) x2/steps counted
Cadence | 2 weeks
  Cadence(steps/min) = steps counted x 60/time(s)
Stride Length | 2 weeks
  SL (m)=Speed(m/s)x cycle time(s)
Pain intensity | 2 weeks
  The numeric pain rating scale is a pain assessment tool that is self-reported or given by a clinician and consists of a numerical point scale with extreme values ranging from "no pain" to "severe pain." O means no pain whereas 10 means severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan